CLINICAL TRIAL: NCT04863040
Title: The Impact of a Classroom-based Physical Activity Breaks on Cognitive Function, Adiposity and Fitness in Preschool Children (MOVI-HIIT)
Brief Title: The Impact of Activity Breaks on Cognitive Function, Adiposity and Fitness in Preschoolers
Acronym: MOVI-HIIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Collaborators: Ministerio de Ciencia e Innovación, Spain (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PID2019-104160RB-I00
Record Dates: First submitted 2021-03-30; First posted 2021-04-28 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Physical Activity; Obesity; Children; Cardiovascular; High Intensity Interval Training; Cognition
Keywords: Physical activity; Obesity; Children; Cognitive function; Academic achievement; Cardiorespiratory fitness; Adiposity; Cardiovascular fitness; Aerobic capacity; High Intensity Interval Training; Preschool
MeSH Terms: conditions — Motor Activity; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual classroom teaching methodology (No Intervention): Students in the CG will receive mandatory lessons on Spain (one 45-minute session of Psychomotor/Physical Education), and the usual classroom teaching methodology. Teachers in the CG schools will be asked not to make any changes to their methodology during the time of the study, with the promise by the research team to share and explain the MOVI-HIIT materials once the interventions are completed.
- Usual classroom teaching methodology + MOVI-HIIT intervention (Experimental): The design of the MOVI-HIIT intervention is framed within the socio-ecological model of behavior modification, in such a way that it will be designed to intervene in the individual, family and school environment. It will have a duration of one school year and will consist of two 5-minute daily physical activity breaks based on intervallic training, five days a week.
  Interventions: Behavioral: MOVI intervention

INTERVENTIONS:
Behavioral: MOVI intervention — Each HIIT break will last approximately 5 minutes and will not require any specific materials. The structure of the HIIT-Rest will be as follows: 1' to describe the work to be done; 3' of work following the HIIT protocol: 6 repetitions of a functional movement such as squats, Jumping Jack or running on site for 10" at high intensity (85-90% of HR max) followed by 20" of recovery (65-75% of HR max); and 1' to perform a return to calm in order to lower the activation and prepare the student body to return to class activities. To increase the workload, and after evaluation of cardiorespiratory capacity, after 12 weeks of program, the HIIT protocol will be changed to 20" of high intensity work alternating with 10" of recovery.
  Other Names: MOVI-HIIT
  Arms: Usual classroom teaching methodology + MOVI-HIIT intervention

SUMMARY:
Project which objective is a) to test the effectiveness, in preschool children, of an integrated physical activity intervention in the classroom based on intervallic training (MOVI-HIIT) on improving executive function, body composition, cardiorespiratory fitness and b) to evaluate teachers' perceptions of barriers and facilitating elements for the implementation and monitoring of MOVI-HIIT interventions in the classroom.

DETAILED DESCRIPTION:
In the last decade, this research group has tested the effectiveness of five interventions in school settings. The first one (MOVI) was carried out in children 8 to 11 years children (4th and 5th year of primary education) and showed a moderate effect in reducing adiposity of schoolchildren with higher body mass index (BMI), and an improvement of the lipid profile without significantly improving the global cardiometabolic risk, because it did not produce a reduction in insulinemia.

The second edition (MOVI-2), carried out with schoolchildren of the same age range, increased the duration and intensity of the sessions, and was focused on the development of muscular strength in order to improve insulinemia levels. The intervention proved to be effective; in addition, data from this intervention showed a modest improvement in girls' aerobic capacity, but not in boys.

The third edition (MOVI-KIDS) was aimed at children aged 4 to 7 years to test the hypotheses that vigorous physical activity at early ages could produce lifelong cardio-metabolic benefits. This study show that, as in the case of the IDEFICS study in children of similar age, the intervention was not effective in improving fitness.

The fourth edition (MOVI-da10!) was carried out at schoolchildren of the same age range, but focusing on active breaks designs, and as a controlled cluster-randomized trial, to test the effectiveness of a classroom-based physical activity intervention on improving, body composition, cardiorespiratory fitness and executive function.

The fifth edition (MOVI-daFit!) was carried out with 9 to 11 years schoolchildren, and consisted in a standardized recreative, non-competitive, physical activity intervention based on games adapted to high intensity interval training methodology (out of school hours, four times by week, one hour session). The aim was to test the effectiveness of an extracurricular physical activity intervention based on high intensity interval training (MOVI-daFit!) on improving cardiorespiratory fitness, cardiometabolic risk, executive function, and academic performance.

The results from these last two editions are currently under process of publishing.

The new edition (MOVI-HIIT) has been designed controlled cluster-randomized trial including 10 schools from Ciudad Real province, Spain. It will include two arms (one intervention and one control arm), in which 5 schools will be randomly assigned to the group in which a physical activity intervention will be performed (MOVI-HIIT), and another 5 schools to the control group in which the usual tasks will be performed.

With the MOVI-HIIT intervention, based on high intensity interval training integrated into the classroom for children of 2nd and 3rd grade of preschool education of one year of duration:

1. Cardiorespiratory fitness (VO2max) will increase in the intervention group (IG) whose values are below the 50th percentile for their age and sex compared to those with the same condition in the control group (CG), with an effect size (standardized mean difference) of 0.3 (moderate). This hypothesis will be used to calculate the sample size in this proposal. Considering only half of schoolchildren with lower cardiorespiratory fitness in IG and CG is due to the fact that VO2 max cannot be increased in trained subjects, and it is possible to increase it very little (less than 2%) in those with acceptable levels of aerobic capacity.
2. It will reduce the percentage of body fat in the IG versus the CG by 6%.
3. It will improve the executive function.

ELIGIBILITY:
Inclusion Criteria:

* Schools in the province of Ciudad Real with at least one class (classroom) at each level (2nd and 3rd of preschool education), and in which the School Board gives its approval to the interventions and to the basal and final evaluations.
* The participating schoolchildren must belong to the 2nd and 3rd year of preschool education, not have any malformation that prevents them from learning the Spanish language (or Spanish sign language), not have any type of physical or mental disorder that parents and/or teachers have identified that prevents the performance of physical activities, not suffer from any chronic disease such as heart disease, diabetes or asthma that, according to the criteria of their pediatrician - after analysis of the program of activities - prevents their participation in them.
* As this is an intervention in the classroom, the school faculty will include the active breaks proposed in the center's programming, for which reason the intervention will be received by all the children in each IG school. However, we will consider school participants to be those who have the consent of the parent or guardian for participation in the study. In addition, schoolchildren must verbally express their willingness to participate in the baseline and final physical examinations.

Exclusion Criteria:

* Children with severe Spanish language learning difficulties.
* Children with serious physical or mental disorders identified by parents or teachers that would impede participation in the programme's activities.
* Children diagnoses of chronic disorders, such as heart disease, diabetes or asthma, which in the opinion of their paediatricians would prevent their participation in the programme's activities (MOVI-HIIT).

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 522 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
VO2max | One year
  Cardiorespiratory fitness, with the Course Navette or 20-m shuttle run test, validated to measure maximum aerobic capacity in children. It will be carried out according to the Léger protocol. This battery adapts the Course Navette test to children under the age of 6.
Executive function | One year
  NIH toolbox battery.
  1. Inhibition/Attention by means of the Flanker Inhibitory Control and Attention test.
  2. Working memory with the List Sorting Working Memory test.
  3. Cognitive flexibility through the DCCS (Dimensional Change Card Sort) test.
Body fat percent | One year
  Body fat percentage measured by Bioimpedance analysis

SECONDARY OUTCOMES:
Health-related quality of life - Parents | One year
  Kiddy-KINDL-R questionnaire version for parents, which has a 0-100 score scale.
Health-related quality of life - Children | One year
  Kiddy-KINDL-R questionnaire version for children, which has a 0-100 score scale.
Mothers' breastfeeding | Baseline measurements
  Parents are going to be ask about what type of feeding had been chosen during their children's first 24 months of life. In each month, systematically, mothers can indicate if their children had been fed by breast milk, artificial milk, both and/or complementary feeding. Mothers can mark one or several options from all those indicated.
Questionnaire ad-hoc about pregnancy | Baseline measurements
  birth weight of their child (Kgr.); maternal weight gain during pregnancy (Kgr.); and parental weight (Kgr.) via direct written questions.
Eating habits | One year
  Children's Eating Habits Questionnaire, which has a 0-30 score scale.
Motor competence | One year
  Movement Assessment Battery for Children - Second Edition (MABC-2). Red zone below 5th percentile which denotes significant movement difficulty; amber zone below or equial to 15th percentile which suggests child at risk of motor problems; green zone, above 15th percentile which indicates no movement problems detected.
Physical activity | One year
  Physical activity will be objectively measured in a subsample of 300 children randomly selected. GENEActive® accelerometers (ActivInsights) will be worn for seven consecutive days, with a fixed frequency of 85.7Hz to collect raw acceleration data measured in "g" for each axis of motion (x,y,z). The data shall be stored directly in the memory of the device and expressed in milli-g units (1000mg =1 g =9.81 m/s2).
Sleep quality | One year
  Sleep quality via acelerometer will be objectively measured in a subsample of 300 children randomly selected. GENEActive® accelerometers (ActivInsights) will be worn for seven consecutive days during nights, with a fixed frequency of 85.7Hz to collect raw acceleration data measured in "g" for each axis of motion (x,y,z). The data shall be stored directly in the memory of the device and expressed in milli-g units (1000mg =1 g =9.81 m/s2).
Energy expenditure from MOVI-HIIIT breaks | One year
  40 schoolchildren of an IG school will be estimated from the oxygen consumption measured with a portable gas analyzer (COSMED® k4b2).
The acute effect of physical exercise on the brain's electrical activity | One year
  40 schoolchildren (20 from the CG and 20 from the IG) will be estimated from the brain activity measured with a portable electroencephalogram (EMOTIV EPOC X).
  14-channel EEG - for whole brain sensing (AF3, AF4, F3, F4, F7, F8, T7, T8, P3, P4, P7, P8, O1, O2)

CONTACTS AND LOCATIONS:
Overall Officials: Mairena Sanchez-Lopez, PhD, Principal Investigator — University of Castilla-La Mancha
Locations (1):
- Social and Health Research Center. Universidad de Castilla-La Mancha, Cuenca, Spain

IPD SHARING:
Plan to Share IPD: No